CLINICAL TRIAL: NCT03442400
Title: A Prospective Study of Fractional Flow Reserve Assessment of Intermediate Coronary Stenoses in Severe Aortic Stenosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: The Cleveland Clinic (Other)
Collaborators: Volcano Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB 17-695
Record Dates: First submitted 2018-02-06; First posted 2018-02-22 (Actual); Results first posted 2023-01-05 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2022-12

CONDITIONS: Coronary Artery Stenoses; Aortic Stenosis
Keywords: Coronary Artery Stenoses; Aortic Stenosis
MeSH Terms: conditions — Coronary Stenosis; Aortic Valve Stenosis

STUDY DESIGN:
Intervention Model Description: A single group of patients with severe aortic stenosis and intermediate coronary stenoses will undergo coronary physiology assessment with iFR/FFR before and after transcatheter aortic valve replacement.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- FFR/iFR arm (Experimental): Volcano iFR/FFR Verrata Plus coronary pressure/flow wire
  Interventions: Device: Volcano iFR/FFR Verrata Plus coronary pressure/flow wire

INTERVENTIONS:
Device: Volcano iFR/FFR Verrata Plus coronary pressure/flow wire — We will measure the degree of flow-limitation of intermediate severity coronary steonses using the iFR/FFR Verrata Plus coronary pressure/flow wire before and after transcatheter aortic valve replacement.

SUMMARY:
Coronary artery blockages can reduce blood flow to the heart muscle. Fractional flow reserve (iFR or FFR) assessment is an invasive tool used to determine how much blood flow is reduced. The investigators will perform iFR/FFR on all intermediate coronary stenoses using standard practice, immediately before (at the time of) transcatheter aortic valve replacement (TAVR) and after successful TAVR. The investigators will compare pre- and post-TAVR iFR/FFR values, and assess short-term outcomes. The investigators hypothesize that iFR/FFR values will be consistently and significantly higher pre-TAVR in comparison with post-TAVR for the same lesions.

DETAILED DESCRIPTION:
The purpose of the study is to determine whether iFR assessment gives a valid assessment of coronary hemodynamics in patients with severe aortic stenosis.

Several factors confound the interpretation of fractional flow reserve (FFR) in patients with severe aortic stenosis (AS) and intermediate severity coronary stenoses, and the widely accepted cut-off value of 0.80 may not be applicable to this patient population. Coronary flow reserve is known to be attenuated under conditions of left ventricular hypertrophy and severe AS, with one study showing improvement in coronary flow reserve after aortic valve replacement. Left ventricular hypertrophy produces fixed resistance secondary to external compression of the coronary microcirculation. This potentially results in failure to achieve maximal hyperemia with adenosine and can lead to false negative FFR results. Neurohormonal influences in aortic stenosis can further attenuate vasodilator response and potentially result in false negative FFR values. Both of these conditions result in the potential deferral of lesions which may have been hemodynamically significant in the absence of severe AS. At present, there are no studies which have demonstrated validity of FFR measurement in patients with severe AS. Here, the investigators propose a prospective study of iFR/FFR in patients with AS and indeterminate coronary lesions undergoing TAVR to understand the hemodynamic consequences of AS on iFR/FFR. The investigators hypothesize that iFR/FFR values will be consistently and significantly higher pre-TAVR in comparison with post-TAVR for the same lesions.

ELIGIBILITY:
Inclusion Criteria:

* All patients who have coronary stenoses between 40-70% severity and who have severe aortic stenosis undergoing TAVR work-up.

Exclusion Criteria:

* Patients with documented intraprocedural hemodynamic instability, shock, or major adverse event (myocardial infarction, aortic rupture/dissection, stroke, left ventricular perforation, cardiac arrest).
* Contraindication to adenosine, presence of cardiogenic shock, presence of acute coronary syndrome.

Ages: 20 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samir R Kapadia, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- The Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FFR/iFR Arm
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | FFR/iFR Arm
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Diabetes [Count of Participants; unit: Participants] | 2
Hypertension [Count of Participants; unit: Participants] | 5
Hyperlipidemia [Count of Participants; unit: Participants] | 5
Kidney disease [Count of Participants; unit: Participants] | 0
Previous percutaneous coronary intervention [Count of Participants; unit: Participants] | 0
Previous MI [Count of Participants; unit: Participants] | 0

OUTCOME MEASURES:

1. Primary Outcome: FFR Values Prior to Transcatheter Aortic Valve Replacement
Description: Hemodynamic significance of a coronary stenosis by measuring FFR immediately prior to TAVR
Time Frame: Immediately prior to transcatheter aortic valve replacement, during the index procedure
Population: 1 patient did not have the FFR value documented
Measure: Mean (Standard Error); unit: ratio
Arm/Group | FFR/iFR Arm
Number analyzed (Participants) | 4
ratio | 0.86 (0.0330088372006)

2. Primary Outcome: FFR Values During the Transcatheter Aortic Valve Replacement (TAVR)
Description: Hemodynamic significance of a coronary stenosis by measuring FFR immediately after TAVR
Time Frame: Immediately after transcatheter aortic valve replacement, during the index procedure
Population: 1 patient did not have the FFR value documented
Measure: Mean (Standard Error); unit: ratio
Arm/Group | FFR/iFR Arm
Number analyzed (Participants) | 4
ratio | 0.91 (0.0335099487715)

ADVERSE EVENTS:
Time Frame: During the index procedure, an average of 1 hour
Groups:
- Interventional Arm: Measure FFR with Volcano Verrata Plus coronary pressure/flow wire during the TAVR procedure.
  By using the Volcano Verrata Plus coronary pressure/flow wire, measure the degree of flow-limitation of intermediate severity coronary steonses using the Verrata Plus coronary pressure/flow wire before and after transcatheter aortic valve replacement.
Arm/Group | Interventional Arm
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2017-05-08): https://cdn.clinicaltrials.gov/large-docs/00/NCT03442400/Prot_001.pdf